CLINICAL TRIAL: NCT05703828
Title: Impact of Chronic Ankle Instability on Gait Loading Strategy
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant professor at faculty of physical therapy, Delta University for Science and Technology
Other Study IDs: Chronic Ankle Instabiility
Record Dates: First submitted 2023-01-08; First posted 2023-01-30 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronic ankle sprain group
- health subjects group

SUMMARY:
compare the dynamic foot print outcomes in subjects suffering from chronic ankle sprain to heathy subjects

ELIGIBILITY:
Inclusion Criteria:

* subjects were suffering from chronic ankle sprain.
* age ranged from 20-30 years old.
* Normal BMI (ranged from 18 to 24.9 Kg/m2)

Exclusion Criteria:

* not suffering from any neuromuscular disorders , deformities

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: use G power soft were
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
loading force | through study completion, an average of 3 months
  force plate form is used to determine foot print parameter e.g. loading force
foot print parameter - ankle rocker | through study completion, an average of 3 months
  force plate form is used to determine foot print parameter ankle rocker

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: Undecided